CLINICAL TRIAL: NCT03416946
Title: A Double-blinded, Randomized, Controlled Trial of Total Knee Replacement Using Custom Cutting Block Instrument vs Regular Instrumentation
Brief Title: Custom Cutting Block Instrument vs Regular Instrumentation Total Knee Replacement (TKR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopaedic Innovation Centre (Other)
Responsible Party: Principal Investigator, Dr. Thomas Turgeon, Orthopaedic Surgeon, Orthopaedic Innovation Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS13322
Record Dates: First submitted 2017-12-13; First posted 2018-01-31 (Actual); Results first posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Osteoarthritis, Knee
Keywords: Total knee replacement
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: The block randomization process will be stratified by surgeon to ensure equal distribution between the two surgical techniques.
Who Masked: Participant
Masking Description: Randomization will occur after enrolment and subjects will be blinded to assignment group. All subjects will be scheduled for and receive the same MRI experience. It is not possible to blind the surgeon to the surgical technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Custom Block Instrumentation (Active Comparator): Patients-specific custom cutting blocks using the Smith and Nephew Visionaire system
  Interventions: Device: Visionaire
- Traditional Instrumentation (Active Comparator): Traditional cutting methods for Total Knee Replacement
  Interventions: Other: Traditional

INTERVENTIONS:
Device: Visionaire — Custom cutting block using MRI to create patient specific instrumentations
  Arms: Custom Block Instrumentation
Other: Traditional — Traditional cutting method
  Arms: Traditional Instrumentation

SUMMARY:
To determine if the use of patient-specific custom cutting blocks for implantation of total knee components results in improved limb alignment and component positioning compared to regular instrumentation.

DETAILED DESCRIPTION:
This is a randomized controlled trial. Patients will be randomized to have their knee implanted using either the patient-specific custom cutting blocks or the regular instrumentation system. Functional and radiographic outcomes will be assessed in a blinded fashion. The Smith and Nephew Legion Primary® total knee system will be used in both groups; this is an implant with a good long term track record based on the Genesis II design. All surgeons have used and are familiar with the regular instrumentation. They will be instructed in the use of the patient-specific custom cutting blocks prior to study initiation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is male or female ages 18 and over.
2. Patient is having primary total knee replacement
3. Patient is willing to sign the informed consent and to come for all study visits.

Exclusion Criteria:

1. Deformity of the femur preventing use of the intra-medullary guide utilized in the regular instrumentation set.
2. Necessity for the use of constrained implants. These types of implants have intra-medullary stems, therefore all bone cuts need to be referenced off intramedullary guides, making image guided bone cuts inappropriate.
3. Patients undergoing knee replacement revision surgery. Theses types of implants also have stems, making the use of image guided bone cuts inappropriate for the same reasons.
4. Patients scheduled for bilateral knee surgery (simultaneous or staged)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Turgeon, MD MPH FRCSC, Principal Investigator — Orthopaedic Innovation Centre
Locations (1):
- Concordia Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turgeon TR, Cameron B, Burnell CD, Hedden DR, Bohm ER. A double-blind randomized controlled trial of total knee replacement using patient-specific cutting block instrumentation versus standard instrumentation. Can J Surg. 2019 Dec 1;62(6):460-467. doi: 10.1503/cjs.018318. PMID 31782643

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Custom Block Instrumentation | Traditional Instrumentation
Started | 25 | 29
Completed | 25 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Custom Block Instrumentation | Traditional Instrumentation | Total
Number analyzed (Participants) | 25 | 29 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (9.2) | 65.7 (9.2) | 64.8 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 40
  Male | 7 | 7 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 25 | 29 | 54
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 33.6 (7.2) | 32.0 (6.0) | 32.76 (6.6)
Knee [Count of Participants; unit: Participants]
  Right | 13 | 12 | 25
  Left | 12 | 17 | 29
Pre-op HKA angle [Mean (Standard Deviation); unit: degree] | -5.2 (5.9) | -6.7 (7.5) | -6.0 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Alignment
Description: Using 3 foot standing film
Time Frame: 8 Weeks
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Custom Block Instrumentation | Traditional Instrumentation
Number analyzed (Participants) | 25 | 29
degree
  Post-op HKA angle | -1.6 (3.2) | -1.8 (2.7)
  Femoral coronal angle | 89.4 (1.9) | 89.3 (2.5)
  Tibial coronal angle | 89.2 (1.5) | 89.1 (1.6)
  Femoral sagittal angle | 87.4 (2.2) | 87.3 (2.7)
  Tibial sagittal angle | 3.8 (3.0) | 7.7 (3.6)
Statistical Analysis 1: Comparison: Custom Block Instrumentation vs Traditional Instrumentation; Test type: Superiority; p = 0.790, t-test, 2 sided — Post-op HKA angle

2. Primary Outcome: Number of HKA Angle Outliers
Description: The angle formed between the mechanical axes of the femur and tibia create the hip-knee-ankle (HKA) angle.
Time Frame: 8 Weeks
Measure: Number; unit: outliers
Arm/Group | Custom Block Instrumentation | Traditional Instrumentation
Number analyzed (Participants) | 25 | 29
outliers | 6 | 10

3. Secondary Outcome: EuroQol (EQ) Five Dimension (5D) Survey
Description: Evaluate change from preoperative baseline to 1 and 2 year post operative in functional outcomes assessments using the EQ-5D (patient reported). The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state, this health state is range from 0 to 1.0. Higher scores indicate improved quality of life within each dimension.
Time Frame: Preoperative, 1 and 2 years
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Custom Block Instrumentation | Traditional Instrumentation
Number analyzed (Participants) | 25 | 29
units on a scale
  Pre-op | 0.760 (0.058) | 0.744 (0.061)
  1 Year | 0.101 (0.090) | 0.110 (0.086)
  2 Years | 0.112 (0.110) | 0.120 (0.098)

4. Secondary Outcome: Oxford Knee Score
Description: Evaluate change from preoperative baseline to 1 and 2 year post operative in functional outcomes assessments using the Oxford 12 scores (patient reported). The score ranges from 0 to 48 with higher scores indicating improved function and less pain.
Time Frame: Preoperative, 1 and 2 years
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Custom Block Instrumentation | Traditional Instrumentation
Number analyzed (Participants) | 25 | 29
units on a scale
  Pre-op | 22.8 (7.8) | 19.6 (6.8)
  Improvement at 1 Year | 10.7 (11.4) | 15.3 (7.7)
  Improvement at 2 Year | 13.3 (12.4) | 12.8 (8.9)

5. Secondary Outcome: Pain Catastrophizing Scale (PCS) Score
Description: Evaluate change from preoperative baseline to 1 and 2 year post operative in functional outcomes assessments using the PCS (patient reported). The total score ranges from 0 to 52 with higher scores indicating greater pain catastrophizing. Sub-scales will not be used in this study.
Time Frame: Preoperative, 1 and 2 years
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Custom Block Instrumentation | Traditional Instrumentation
Number analyzed (Participants) | 25 | 29
units on a scale
  Pre-op | 14.0 (12.3) | 17.4 (11.9)
  Improvement at 1 Year | 9.1 (12.3) | 10.5 (14.4)
  Improvement at 2 Year | 8.0 (13.7) | 6.4 (14.9)

6. Secondary Outcome: Hip Pain
Description: Evaluate change from preoperative baseline to 1 and 2 year post operative in functional outcomes assessments using the Pain Visual Analog Scale (VAS). The scale is from 0 to 100, 0=no pain and at 100= worst pain. (patient reported).
Time Frame: Preoperative, 1 and 2 years
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Custom Block Instrumentation | Traditional Instrumentation
Number analyzed (Participants) | 25 | 29
units on a scale
  Pre-op | 61.6 (23.4) | 67.4 (20.6)
  Improvement at 1 Year | -38.4 (34.4) | -40.1 (32.9)
  Improvement at 2 Year | -40.8 (40.1) | -46.3 (24.2)

7. Secondary Outcome: University of California Los Angeles (UCLA) Activity Score
Description: Evaluate change from preoperative baseline to 1 and 2 year post operative in activity level assessments using the UCLA Activity score (patient reported). The scale ranges from 1-10 with higher values associated with more intense activities.
Time Frame: Preoperative, 1 and 2 years
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Custom Block Instrumentation | Traditional Instrumentation
Number analyzed (Participants) | 25 | 29
units on a scale
  Pre-op | 4.4 (1.8) | 3.4 (1.1)
  Improvement at 1 Year | 0.8 (1.92) | 1.6 (1.6)
  Improvement at 2 Year | 1.0 (2.0) | 1.6 (1.7)

8. Secondary Outcome: Patient Satisfaction
Description: Evaluate change from preoperative baseline to 1 and 2 year post operative in functional outcomes assessments using the Satisfaction Visual Analog Scale (VAS). The scale is from 0 to 100, 0=Not Satisfied and at 100=Satisfied. (patient reported).
Time Frame: Preoperative, 1 and 2 years
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Custom Block Instrumentation | Traditional Instrumentation
Number analyzed (Participants) | 25 | 29
units on a scale
  Pre-op | 23.0 (23.5) | 25.6 (26.2)
  Improvement at 1 Year | 59.1 (31.6) | 57.4 (28.5)
  Improvement at 2 Year | 62.0 (31.3) | 56.0 (29.6)

9. Other Pre Specified Outcome: Other Measure: Time
Description: Surgical and tourniquet time
Time Frame: Intra-operative
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Custom Block Instrumentation | Traditional Instrumentation
Number analyzed (Participants) | 25 | 29
Minutes | 64.2 (16.5) | 57 (14)

10. Other Pre Specified Outcome: Blood Loss
Description: Blood loss during surgery >100ml (n)
Time Frame: Intra-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Custom Block Instrumentation | Traditional Instrumentation
Number analyzed (Participants) | 25 | 29
Participants | 5 | 10

11. Other Pre Specified Outcome: Length of Stay (LOS)
Description: Length of hospital stay
Time Frame: Peri-operative
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Custom Block Instrumentation | Traditional Instrumentation
Number analyzed (Participants) | 25 | 29
Days | 4.0 (1.5) | 4.2 (2.6)

12. Other Pre Specified Outcome: Other Measures: Adverse Events
Description: Peri-operative complications such as deep venous thrombosis, pulmonary emboli, wound complications and cardiac events.
  Post-operative complication such as infection, loosening, etc.
Time Frame: Peri-operative, intra-operative and post-operative
Measure: Number; unit: participants
Arm/Group | Custom Block Instrumentation | Traditional Instrumentation
Number analyzed (Participants) | 25 | 29
participants | 4 | 1

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | Custom Block Instrumentation | Traditional Instrumentation
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/29
Serious Adverse Events (participants affected / at risk) | 4/25 | 1/29
Other Adverse Events (participants affected / at risk) | 0/25 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Custom Block Instrumentation (N=25) | Traditional Instrumentation (N=29)
Revision (Infections and infestations) | 2 (2) | 0 (0) — Patient required revision surgery of the knee due to infection.
Revision (Surgical and medical procedures) | 0 (0) | 1 (1) — Patient required revision surgery due to pain of unknown origin.
Revision (Surgical and medical procedures) | 1 (1) | 0 (0) — Patient required revision surgery due to an accident
Manipulation (Surgical and medical procedures) | 1 (1) | 0 (0) — Patient required knee manipulation under anesthesia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-06-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT03416946/Prot_SAP_000.pdf